CLINICAL TRIAL: NCT04853368
Title: A Phase 2 Study of Galicaftor/Navocaftor/ABBV-119 or Galicaftor/Navocaftor/ABBV-576 Combination Therapies in Subjects With Cystic Fibrosis Who Are Homozygous or Heterozygous for the F508del Mutation
Brief Title: Study to Evaluate Adverse Events and Change in Disease Activity With Oral Capsules of Galicaftor/Navocaftor/ABBV-119 or Galicaftor/Navocaftor/ABBV-576 Combination Therapies in Adult Participants With Cystic Fibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M19-771; 2020-005805-25 (EudraCT Number)
Record Dates: First submitted 2021-04-19; First posted 2021-04-21 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Cystic Fibrosis (CF)
Keywords: Cystic Fibrosis (CF); Galicaftor; Navocaftor; ABBV-119; ABBV-576
MeSH Terms: conditions — Cystic Fibrosis | interventions — GLPG2222

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- F508del Homozygous Cystic Fibrosis (CF) Participants (Experimental): F508del homozygous cystic fibrosis (CF) participants receive galicaftor/navocaftor dual combination (28 days) followed by galicaftor/navocaftor/ABBV-119 triple combination therapy (28 days).
  Interventions: Drug: Galicaftor; Drug: Navocaftor; Drug: ABBV-119
- F508del Heterozygous CF Participants (Active Drug Group) (Experimental): F508del heterozygous CF participants receive galicaftor/navocaftor/ABBV-119 combination therapy (28 days).
  Interventions: Drug: Galicaftor; Drug: Navocaftor; Drug: ABBV-119
- F508del Heterozygous CF Participants (Placebo Group) (Placebo Comparator): F508del heterozygous CF participants receive placebo (28 days).
  Interventions: Drug: Placebo
- F508del Homozygous and Heterozygous CF Participants (Experimental): F508del homozygous and heterozygous CF participants receive galicaftor/navocaftor/ABBV-576 triple combination therapy for 28 days.
  Interventions: Drug: ABBV-576; Drug: Galicaftor; Drug: Navocaftor

INTERVENTIONS:
Drug: ABBV-576 — Oral capsules
  Arms: F508del Homozygous and Heterozygous CF Participants
Drug: Galicaftor — Oral capsules
  Other Names: ABBV-2222
  Arms: F508del Heterozygous CF Participants (Active Drug Group); F508del Homozygous Cystic Fibrosis (CF) Participants; F508del Homozygous and Heterozygous CF Participants
Drug: Placebo — Oral capsules
  Arms: F508del Heterozygous CF Participants (Placebo Group)
Drug: Navocaftor — Oral capsules
  Other Names: ABBV-3067
  Arms: F508del Heterozygous CF Participants (Active Drug Group); F508del Homozygous Cystic Fibrosis (CF) Participants; F508del Homozygous and Heterozygous CF Participants
Drug: ABBV-119 — Oral capsules
  Arms: F508del Heterozygous CF Participants (Active Drug Group); F508del Homozygous Cystic Fibrosis (CF) Participants

SUMMARY:
Cystic Fibrosis (CF) is a rare, life-threatening, genetic disease that affects the lungs and digestive system, significantly impairing the quality of life, with those affected having a median age of death at 40. The main objective of this study is to assess how safe and effective is the combination therapy of galicaftor/navocaftor/ABBV-119 or Galicaftor/Navocaftor/ABBV-576 in adult participants with CF who are homozygous or heterozygous for the F508del mutation in each arm.

Galicaftor/Navocaftor/ABBV-119 combination therapy and Galicaftor/Navocaftor/ABBV-576 is being developed as an investigational drug for the treatment of CF. Study doctors place participants in 1 of the 4 groups, called treatment arms. Each group receives a different treatment. Around 90 adult participants with a diagnosis of CF will be enrolled in the study around approximately 35 sites worldwide.

Participants in arm 1 will receive oral capsules of galicaftor/navocaftor dual combination for 28 days followed by galicaftor/navocaftor/ABBV-119 triple combination for 28 days. Participants in arms 2 and 3 will receive the galicaftor/navocaftor/ABBV-119 triple combination or placebo for 28 days. Participants in arm 4 will receive galicaftor/navocaftor/ABBV-576 triple combination therapy for 28 days. For all study arms, ABBV-576, galicaftor, navocaftor, will be given once daily and ABBV-119 twice a day.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

DETAILED DESCRIPTION:
Participants in Cohorts 1 and 3 will receive Open-label therapy. Participants in Cohorts 2 will receive Double-blinded therapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical diagnosis of cystic fibrosis (CF).
* Arm 1 participants with genotype homozygous for the F508del CF transmembrane conductance regulator (CFTR) mutation and not receiving elexacaftor/tezacaftor/ivacaftor (ETI) treatment .
* Arm 2 and 3 participants with genotype heterozygous for the F508del CFTR mutation and a minimal function mutation and not receiving ETI treatment.
* Arm 4 participants with genotype either homozygous or heterozygous for the F508del mutation. Participants must be receiving stable ETI treatment.
* Percent predicted forced expiratory volume in 1 second (ppFEV1) >= 40% and <=90% of predicted normal for age, gender and height at screening.
* For arms 1 and 2: sweat chloride (SwCl) >= 60 mmol/L at screening. For participants who participated in Study M19-530, it is acceptable to use a SwCl value that the central lab provided in Study M19-530 to establish eligibility.
* Weight >= 35 kg at screening and Day -28 for arm 1 or day 1 for arms 2 to 4.

Exclusion Criteria:

- Clinically significant laboratory values at screening that would pose undue risk for the participant or interfere with safety assessments (per the investigator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (41):
- United States (22):
  - Velocity Clinical Research /ID# 248675, Mobile, Alabama
  - University of Southern California /ID# 249147, Los Angeles, California
  - Ventura County Medical Center /ID# 248586, Ventura, California
  - Central FL Pulmonary Orlando /ID# 245432, Orlando, Florida
  - University of Kansas Health Sy /ID# 249056, Kansas City, Kansas
  - Boston Children's Hospital /ID# 248646, Boston, Massachusetts
  - Harper University Hospital /ID# 248917, Detroit, Michigan
  - Washington University-School of Medicine /ID# 245393, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center /ID# 245706, Lebanon, New Hampshire
  - Dartmouth Hitchcock Manchester /ID# 248795, Manchester, New Hampshire
  - Albany Medical College-Pulmonary /ID# 248838, Albany, New York
  - Northwell Health/Long Island Jewish Hospital /ID# 248916, New Hyde Park, New York
  - New York Medical College /ID# 248640, Valhalla, New York
  - UH Cleveland Medical Center /ID# 245433, Cleveland, Ohio
  - ProMedica Toledo Harris McIntosh /ID# 248627, Toledo, Ohio
  - University of Oklahoma HSC /ID# 249190, Oklahoma City, Oklahoma
  - Penn State Health /ID# 248585, Hershey, Pennsylvania
  - Medical University of South Carolina /ID# 245403, Charleston, South Carolina
  - Vanderbilt University Medical Center /ID# 245400, Nashville, Tennessee
  - The Univ Texas HSC at Tyler /ID# 248498, Tyler, Texas
  - Children's Hospital of Richmond at VCU /ID# 248561, Richmond, Virginia
  - Medical College of Wisconsin - Plank Rd /ID# 249079, Milwaukee, Wisconsin
- Australia (7):
  - Royal Prince Alfred Hospital /ID# 228781, Camperdown, New South Wales
  - Westmead Hospital /ID# 227281, Westmead, New South Wales
  - Mater Misericordiae Limited /ID# 227279, South Brisbane, Queensland
  - Royal Adelaide Hospital /ID# 228486, Adelaide, South Australia
  - Alfred Health /ID# 227283, Melbourne, Victoria
  - Royal Children's Hospital /ID# 227280, Parkville, Victoria
  - Institute for Respiratory Health /ID# 227624, Nedlands, Western Australia
- Belgium (4):
  - Uza /Id# 228533, Edegem, Antwerpen
  - UZ Brussel /ID# 226607, Jette, Brussels Capital
  - UZ Gent /ID# 226605, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 226608, Leuven, Vlaams-Brabant
- Orszagos Koranyi Pulmonologiai Intezet /ID# 228810, Budapest, Hungary
- Netherlands (3):
  - Erasmus Medisch Centrum /ID# 234254, Rotterdam, South Holland
  - Academisch Medisch Centrum /ID# 234253, Amsterdam
  - HagaZiekenhuis /ID# 234138, The Hague
- New Zealand (2):
  - Greenlane Clinical Centre /ID# 227282, Epsom, Auckland
  - Christchurch Hospital /ID# 227335, Christchurch, Canterbury
- Slovakia (2):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica /ID# 228044, Banská Bystrica
  - Univerzitna nemocnica Bratislava Nemocnica Ruzinov /ID# 228042, Bratislava

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this 2-part study, Cystic Fibrosis (CF) participants either homozygous or heterozygous for F508del mutation were placed in cohorts based on genotype and treatment status of ETI therapy. In Part 1, Cohort 1(Day -29 to -1) (C1) completed Galicaftor + Navocaftor (G+N) dual combination therapy for 28 days (d) and automatically started Part 2. In Part 2, C1(d1 - 29) and C2(d1 - 29) received G+N+ABBV-119 triple combination, and C3(d1 -29) received G+N+ABBV-576 triple combination for 28d
Groups:
- C1(d-29 to -1) Dual Combo G + N: F508del Homozygous cystic fibrosis (CF) participants received Galicaftor/ Navocaftor dual combination (Day -29 to -1).
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
- C1(d1 - 29) Triple Combo G + N + ABBV-119: F508del homozygous CF participants from Cohort 1(Day -29 to -1) who received G + N dual combination therapy
  followed by
  Galicaftor/Navocaftor/ABBV-119 triple combination therapy (Day 1- 29).
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
  ABBV-119: 210 mg BID, Oral capsules
- C2(d1 - 29) Triple Combo G + N + ABBV-119: F508del Heterozygous CF participants received Galicaftor/Navocaftor/ABBV-119 triple combination therapy (Day 1 - 29).
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
  ABBV-119: 210 mg BID, Oral capsules
- C2(d1 - 29) Placebo: F508del Heterozygous CF participants received placebo (Day 1 - 29).
  Placebo: Oral capsules
- C3 (d1 - 29) Triple Combo G + N + ABBV-576 for F508del Homo: F508del Homozygous CF participants received Galicaftor/Navocaftor/ABBV-576 triple combination therapy (Day 1 - 29).
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
  ABBV-576: 5 mg QD, Oral capsules
- C3 (d1 - 29) Triple Combo G + N + ABBV-576 for F508del Hetero: F508del Heterozygous CF participants received Galicaftor/Navocaftor/ABBV-576 triple combination therapy (Day 1 - 29).
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
  ABBV-576: 5 mg QD, Oral capsules
Period: Part 1 (Day -29 to -1)
Arm/Group | C1(d-29 to -1) Dual Combo G + N | C1(d1 - 29) Triple Combo G + N + ABBV-119 | C2(d1 - 29) Triple Combo G + N + ABBV-119 | C2(d1 - 29) Placebo | C3 (d1 - 29) Triple Combo G + N + ABBV-576 for F508del Homo | C3 (d1 - 29) Triple Combo G + N + ABBV-576 for F508del Hetero
Started | 24 | 0 | 0 | 0 | 0 | 0
Completed | 24 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (Day 1-29)
Arm/Group | C1(d-29 to -1) Dual Combo G + N | C1(d1 - 29) Triple Combo G + N + ABBV-119 | C2(d1 - 29) Triple Combo G + N + ABBV-119 | C2(d1 - 29) Placebo | C3 (d1 - 29) Triple Combo G + N + ABBV-576 for F508del Homo | C3 (d1 - 29) Triple Combo G + N + ABBV-576 for F508del Hetero
Started | 0 | 24 | 9 | 4 | 9 | 2
Completed | 0 | 22 | 9 | 4 | 8 | 2
Not Completed | 0 | 2 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) includes all enrolled subjects (randomized subjects for Cohort 2) who received at least 1 dose of study drug as dual or triple combination (or corresponding placebo). The FAS was used for demographics and baseline characteristics analyses.
Groups:
- C1 (d -29 to -1) Dual Combo: G + N, and C1 (d1 - 29) Triple Combo: G + N + ABBV-119 for F508del Homo: Cohort 1 (Day -29 to -1):
  F508del Homozygous cystic fibrosis (CF) participants received Galicaftor/Navocaftor dual combination therapy:
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
  Cohort 1 (Day 1 to 29):
  F508del Homozygous cystic fibrosis CF participants from Cohort 1 (Day -29 to -2) dual combination who received Galicaftor/Navocaftor dual combination followed by Galicaftor/Navocaftor/ABBV-119 triple combination therapy:
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
  ABBV-119: 210 mg BID, Oral capsules
- Cohort 2 (d1 - 29) Triple Combo: G + N + ABBV-119 for F508del Heterozygous: F508del Heterozygous CF participants received Galicaftor/Navocaftor/ABBV-119 triple combination therapy(Day 1 - 29).
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
  ABBV-119: 210 mg BID, Oral capsules
- Cohort 2 (d1 - 29) Placebo for F508del Heterozygous: F508del Heterozygous CF participants received placebo (Day 1 - 29).
  Placebo: Oral capsules
- Cohort 3 (d1 - 29) Triple Combo: G + N + ABBV-576 for F508del Homozygous: F508del Homozygous CF participants receive Galicaftor/Navocaftor/ABBV-576 triple combination therapy (Day 1 - 29).
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
  ABBV-576: 5 mg QD, Oral capsules
- Cohort 3 (d1 - 29) Triple Combo: G + N + ABBV-576 for F508del Heterozygous: F508del Heterozygous CF participants received Galicaftor/nNavocaftor/ABBV-576 triple combination therapy (Day 1 - 29).
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
  ABBV-576: 5 mg QD, Oral capsules
- Total: Total of all reporting groups
Arm/Group | C1 (d -29 to -1) Dual Combo: G + N, and C1 (d1 - 29) Triple Combo: G + N + ABBV-119 for F508del Homo | Cohort 2 (d1 - 29) Triple Combo: G + N + ABBV-119 for F508del Heterozygous | Cohort 2 (d1 - 29) Placebo for F508del Heterozygous | Cohort 3 (d1 - 29) Triple Combo: G + N + ABBV-576 for F508del Homozygous | Cohort 3 (d1 - 29) Triple Combo: G + N + ABBV-576 for F508del Heterozygous | Total
Number analyzed (Participants) | 24 | 9 | 4 | 9 | 2 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 9 | 4 | 9 | 2 | 48
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 1 | 2 | 2 | 17
  Male | 15 | 6 | 3 | 7 | 0 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 24 | 9 | 4 | 9 | 1 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 24 | 8 | 4 | 9 | 2 | 47
  More than one race | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 8 | 5 | 2 | 1 | 0 | 16
  Hungary | 6 | 1 | 0 | 0 | 0 | 7
  Netherlands | 1 | 1 | 1 | 0 | 0 | 3
  New Zealand | 5 | 2 | 1 | 0 | 0 | 8
  Slovakia | 4 | 0 | 0 | 0 | 0 | 4
  United States | 0 | 0 | 0 | 8 | 2 | 10
Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) (%) at Baseline (Day 1) [Mean (Standard Deviation); unit: percent predicted FEV1 (%)] — Note: Percentages calculated on non-missing/non-unknown values. @ Baseline refers to (1) the last value before the first dose of the Dual Therapy for the Cohort 1 dual run-in summary, (2) the last value before the first dose of the Triple Therapy or matching placebo for the other summaries.
  & Subjects may have more than one microbiology history in the past year. Percentages were calculated based on N. Population: The number of participants analyzed for each Cohort varied from Overall analyzed as follows: Cohort 1 (N=24); Cohort 2 (N=13); Cohort 3 (N=11).
  percent predicted FEV1 (%)
    Cohort 1 (Day 1 - 29): number analyzed (Participants) | 24 | 0 | 0 | 0 | 0 | 24
    Cohort 1 (Day 1 - 29) | 57.0 (14.63) |  |  |  |  | 57.0 (14.63)
    Cohort 2 (Day 1 - 29): number analyzed (Participants) | 0 | 9 | 4 | 0 | 0 | 13
    Cohort 2 (Day 1 - 29) |  | 62.9 (18.27) | 67.3 (19.97) |  |  | 64.2 (18.07)
    Cohort 3 (Day 1 - 29): number analyzed (Participants) | 0 | 0 | 0 | 9 | 2 | 11
    Cohort 3 (Day 1 - 29) |  |  |  | 57.0 (19.77) | 51.0 (5.66) | 55.9 (17.94)
Sweat Chloride (SwCl) in mmol/L at Baseline (Day 1) Cohort 3 [Mean (Standard Deviation); unit: mmol/L] — Note: @ Baseline refers to the last value before the first dose of the triple combination therapy.
  * The genotype information is based on the central lab test result. When this information is not available, the CFTR genotype documented at the screening visit is used. Population: The number of participants analyzed for each Cohort varied from Overall analyzed as follows: Cohort 1 (N=24); Cohort 2 (N=13); Cohort 3 (N=11).
  mmol/L
    Cohort 3 (Day 1 - 29): number analyzed (Participants) | 0 | 0 | 0 | 9 | 2 | 11
    Cohort 3 (Day 1 - 29) |  |  |  | 42.94 (10.333) | 26.50 (4.950) | 39.95 (11.494)
    Cohort 1 (Day 1 - 29): number analyzed (Participants) | 24 | 0 | 0 | 0 | 0 | 24
    Cohort 1 (Day 1 - 29) | 76.71 (13.127) |  |  |  |  | 76.71 (13.127)
    Cohort 2 (Day1 - 29): number analyzed (Participants) | 0 | 9 | 4 | 0 | 0 | 13
    Cohort 2 (Day1 - 29) |  | 93.61 (12.437) | 98.38 (9.978) |  |  | 95.08 (11.543)

OUTCOME MEASURES:

1. Primary Outcome: Cohorts 1 and 2: Absolute Change From Baseline Through Day 29 in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration and is used as a measure of lung function. Mixed-effect model with repeated measures (MMRM) was used for the analyses.
Time Frame: Day 1 (Baseline) through Day 29
Population: The Per-Protocol (PP) Population includes all enrolled subjects (randomized subjects for Cohort 2) who carry the intended CFTR mutation based on central lab report and received at least one dose of the Triple Therapy or placebo.
Measure: Mean (Standard Deviation); unit: percent predicted FEV1 (%ppFEV1)
Groups:
- Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous: F508del homozygous CF participants from Cohort 1(Day -29 to -1) who received Galicaftor/Navocaftor dual combination therapy
  followed by
  Galicaftor/Navocaftor/ABBV-119 triple combination therapy (Day 1- 29).
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
  ABBV-119: 210 mg BID, Oral capsules
- Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous: F508del Heterozygous CF participants received Galicaftor/Navocaftor/ABBV-119 triple combination therapy (Day 1 - 29).
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
  ABBV-119: 210 mg BID, Oral capsules
- Cohort 2 (Day 1 - 29) Placebo for F508del Heterozygous: F508del Heterozygous CF participants received placebo (Day 1 - 29).
  Placebo: Oral capsules
Arm/Group | Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous | Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous | Cohort 2 (Day 1 - 29) Placebo for F508del Heterozygous
Number analyzed (Participants) | 20 | 7 | 4
percent predicted FEV1 (%ppFEV1) | 2.2 (3.68) | 2.6 (5.62) | -2.0 (6.63)
Statistical Analysis 1: Comparison: Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous; Test type: Superiority; p = 0.002, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; Primary analysis of ppFEV1 using MMRM excludes data inconsistent with baseline in terms of the timing of bronchodilator or airway clearance regimen; LS Mean of Difference = 2.6, 90% CI 2-sided [1.22 to 4.04], Standard Error of Mean 0.84
Statistical Analysis 2: Comparison: Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous; Test type: Superiority; p = 0.254, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; [statistical method as in outcome 1, analysis 1]; LS Mean of Difference = 1.3, 90% CI 2-sided [-2.07 to 4.67], Standard Error of Mean 1.92
Statistical Analysis 3: Comparison: Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous vs Cohort 2 (Day 1 - 29) Placebo for F508del Heterozygous; Test type: Superiority; p = 0.402, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; [statistical method as in outcome 1, analysis 1]; LS Mean of Difference = 0.9, 90% CI 2-sided [-5.07 to 6.77]

2. Primary Outcome: Cohort 3: Absolute Change From Baseline Through Day 29 in Sweat Chloride (SwCl) in mmol/L
Description: Sweat collection was performed to evaluate sweat chloride concentration. SwCl is a biomarker of cystic fibrosis transmembrane conductance regulator (CFTR) activity. Persons with CF have higher levels of chloride in their sweat. MMRM was used for the analysis.
Time Frame: Day 1 (Baseline) through Day 29
Population: as for outcome 1
Measure: Mean (Full Range); unit: Milli-mole/Liter (mmol/L)
Groups:
- Cohort 3 (Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Homozygous: F508del Homozygous CF participants received Galicaftor/Navocaftor/ABBV-576 triple combination therapy (Day 1 - 29).
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
  ABBV-576: 5 mg QD, Oral capsules
- Cohort 3 (Day 1 - 29)Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Heterozygous: F508del Heterozygous CF participants received Galicaftor/Navocaftor/ABBV-576 triple combination therapy (Day 1 - 29).
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
  ABBV-576: 5 mg QD, Oral capsules
Arm/Group | Cohort 3 (Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Homozygous | Cohort 3 (Day 1 - 29)Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Heterozygous
Number analyzed (Participants) | 1 | 1
Milli-mole/Liter (mmol/L) | 24 [24 to 24] | 40 [40 to 40]

3. Secondary Outcome: Cohorts 1 and 2: Absolute Change From Baseline Through Day 29 in Sweat Chloride (SwCl) in mmol/L
Description: Sweat collection was performed to evaluate sweat chloride concentration. SwCl is a biomarker of CFTR activity. Persons with CF have higher levels of chloride in their sweat. MMRM was used for the analysis.
Time Frame: Day 1 (Baseline) through Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous | Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous | Cohort 2 (Day 1 - 29) Placebo for F508del Heterozygous
Number analyzed (Participants) | 20 | 7 | 4
mmol/L | 5.7 (10.78) | -11.5 (16.61) | 2.5 (4.56)
Statistical Analysis 1: Comparison: Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous; Test type: Superiority; p = 0.022, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; The LS mean is estimated using the mixed-Effect model repeat measurement method; LS Mean of Difference = 5.5, 90% CI 2-sided [1.07 to 9.92], Standard Error of Mean 2.63
Statistical Analysis 2: Comparison: Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous vs Cohort 2 (Day 1 - 29) Placebo for F508del Heterozygous; Test type: Superiority; p = 0.043, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; The LS mean is estimated using the mixed-Effect model repeat measurement method; LS Mean of Difference = -14.1, 90% CI 2-sided [-27.59 to -0.62]

4. Secondary Outcome: Absolute Change From Baseline Through Day 29 in Forced Vital Capacity (FVC)
Description: FVC is the total amount of air exhaled during forced expiratory volume (FEV) test and is a lung function test that is measured during spirometry. MMRM was used for the analyses.
Time Frame: Day 1 (Baseline) through Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters (L)
Groups:
- Cohort 3(Day 1 - 29)Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Heterozygous: F508del Heterozygous CF participants received Galicaftor/nNavocaftor/ABBV-576 triple combination therapy (Day 1 - 29).
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
  ABBV-576: 5 mg QD, Oral capsules
Arm/Group | Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous | Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous | Cohort 2 (Day 1 - 29) Placebo for F508del Heterozygous | Cohort 3 (Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Homozygous | Cohort 3(Day 1 - 29)Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Heterozygous
Number analyzed (Participants) | 20 | 7 | 4 | 3 | 1
Liters (L) | 0.10 (0.256) | 0.05 (0.269) | -0.07 (0.297) | -0.22 (0.318) | -0.28 (NA) — Not applicable; value could not be estimated due to n=1
Statistical Analysis 1: Comparison: Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous; Test type: Superiority; p = 0.003, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; The LS mean is estimated using the mixed-Effect model repeat measurement method; LS Mean of Difference = 0.14, 90% CI 2-sided [0.059 to 0.219], Standard Error of Mean 0.047
Statistical Analysis 2: Comparison: Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous; Test type: Superiority; p = 0.475, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; The LS mean is estimated using the mixed-Effect model repeat measurement method; LS Mean of Difference = -0.01, 90% CI 2-sided [-0.162 to 0.150], Standard Error of Mean 0.089
Statistical Analysis 3: Comparison: Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous vs Cohort 2 (Day 1 - 29) Placebo for F508del Heterozygous; Cohort 2: Difference between Triple Therapy and Placebo; Test type: Superiority; p = 0.352, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; The LS mean is estimated using the mixed-Effect model repeat measurement method; LS Mean of Difference = -0.06, 90% CI 2-sided [-0.332 to 0.212]

5. Secondary Outcome: Absolute Change From Baseline Through Day 29 in Forced Expiratory Flow at Mid-Lung Capacity (FEF25-75)
Description: FEF25-75 is a lung function test that is measured during spirometry, and is defined as the forced expiratory flow between 25% and 75% of vital capacity (mid-lung capacity). MMRM was used for analyses.
Time Frame: Day 1 (Baseline) through Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters/second (L/sec)
Groups:
- Cohort 2 (Day 1 - 29) Placebo F508del Heterozygous: F508del Heterozygous CF participants received placebo (Day 1 - 29).
  Placebo: Oral capsules
- Cohort 3 (Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Homozygous: F508del Homozygous CF participants receive Galicaftor/Navocaftor/ABBV-576 triple combination therapy (Day 1 - 29).
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
  ABBV-576: 5 mg QD, Oral capsules
Arm/Group | Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous | Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous | Cohort 2 (Day 1 - 29) Placebo F508del Heterozygous | Cohort 3 (Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Homozygous | Cohort 3(Day 1 - 29)Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Heterozygous
Number analyzed (Participants) | 20 | 7 | 4 | 3 | 1
Liters/second (L/sec) | 0.067 (0.2038) | 0.134 (0.2506) | -0.082 (0.1947) | -0.329 (0.378) | -0.263 (NA) — Not applicable; value could not be estimated due to n=1
Statistical Analysis 1: Comparison: Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous; Test type: Superiority; p = 0.017, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; The LS mean is estimated using the mixed-Effect model repeat measurement method; LS Mean of Difference = 0.089, 90% CI 2-sided [0.0209 to 0.1568], Standard Error of Mean 0.0403
Statistical Analysis 2: Comparison: Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous; Test type: Superiority; p = 0.169, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; The LS mean is estimated using the mixed-Effect model repeat measurement method; LS Mean of Difference = 0.103, 90% CI 2-sided [-0.1814 to 0.2880], Standard Error of Mean 0.1033
Statistical Analysis 3: Comparison: Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous vs Cohort 2 (Day 1 - 29) Placebo F508del Heterozygous; Test type: Superiority; p = 0.230, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; The LS mean is estimated using the mixed-Effect model repeat measurement method; Mean Difference (Final Values) = 0.136, 90% CI 2-sided [-0.1809 to 0.4527]

6. Secondary Outcome: Relative Changes From Baseline Through Day 29 in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration and is used as a measure of lung function. MMRM was used for the analyses. Note: The primary analysis of ppFEV1 using MMRM excludes data that are inconsistent with baseline in terms of the timing of bronchodilator or airway clearance regimen.
Time Frame: Day 1 (Baseline) through Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % ppFEV1
Arm/Group | Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous | Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous | Cohort 2 (Day 1 - 29) Placebo F508del Heterozygous | Cohort 3 (Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Homozygous | Cohort 3(Day 1 - 29)Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Heterozygous
Number analyzed (Participants) | 20 | 7 | 4 | 3 | 1
% ppFEV1 | 3.8 (6.07) | 3.3 (8.15) | -4.9 (12.25) | -9.1 (5.12) | -19.1 (NA) — value could not be estimated due to n=1
Statistical Analysis 1: Comparison: Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous; Test type: Superiority; p = 0.002, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; LS Mean of Difference = 4.4, 90% CI 2-sided [2.04 to 6.78]
Statistical Analysis 2: Comparison: Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous; Test type: Superiority; p = 0.350, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; LS Mean of Difference = 1.3, 90% CI 2-sided [-4.42 to 6.97]
Statistical Analysis 3: Comparison: Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous vs Cohort 2 (Day 1 - 29) Placebo F508del Heterozygous; Test type: Superiority; p = 0.412, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; LS Mean of Difference = 1.3, 90% CI 2-sided [-8.75 to 11.34]

7. Secondary Outcome: Relative Changes From Baseline Through Day 29 in Forced Vital Capacity (FVC)
Description: FVC is the total amount of air exhaled during FEV test and is a lung function test that is measured during spirometry. MMRM was used for the analyses.
Time Frame: Day 1 (Baseline) through Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters (L)
Groups:
- Cohort 3 (Day 1 - 29)Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Homozygous: F508del Homozygous CF participants receive Galicaftor/Navocaftor/ABBV-576 triple combination therapy (Day 1 - 29).
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
  ABBV-576: 5 mg QD, Oral capsules
- Cohort 3(Day 1 - 29)Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Heterozygous: F508del Heterozygous CF participants received Galicaftor/Navocaftor/ABBV-576 triple combination therapy (Day 1 - 29).
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
  ABBV-576: 5 mg QD, Oral capsules
Arm/Group | Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous | Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous | Cohort 2 (Day 1 - 29) Placebo for F508del Heterozygous | Cohort 3 (Day 1 - 29)Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Homozygous | Cohort 3(Day 1 - 29)Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Heterozygous
Number analyzed (Participants) | 20 | 7 | 4 | 3 | 1
Liters (L) | 3.75 (7.006) | 1.07 (6.524) | -2.06 (8.004) | -6.01 (8.782) | -16.91 (NA) — value could not be estimated due to n=1
Statistical Analysis 1: Comparison: Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous; Test type: Superiority; p < 0.001, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; LS Mean of Difference = 4.36, 90% CI 2-sided [2.190 to 6.524]
Statistical Analysis 2: Comparison: Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous; Test type: Superiority; p = 0.396, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; LS Mean of Difference = -0.59, 90% CI 2-sided [-4.449 to 3.268]
Statistical Analysis 3: Comparison: Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous vs Cohort 2 (Day 1 - 29) Placebo for F508del Heterozygous; Test type: Superiority; p = 0.305, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; LS Mean of Difference = -2.00, 90% CI 2-sided [-8.724 to 4.732]

8. Secondary Outcome: Relative Changes From Baseline Through Day 29 in Forced Expiratory Flow at Mid-Lung Capacity (FEF25-75)
Description: as for outcome 5
Time Frame: Day 1 (Baseline) through Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters/second (L/sec)
Arm/Group | Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous | Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous | Cohort 2 (Day 1 - 29) Placebo for F508del Heterozygous | Cohort 3 (Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Homozygous | Cohort 3(Day 1 - 29)Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Heterozygous
Number analyzed (Participants) | 20 | 7 | 4 | 3 | 1
Liters/second (L/sec) | 4.553 (13.2453) | 8.701 (12.9781) | -6.449 (25.1954) | -8.288 (24.409) | -25.784 (NA) — value could not be estimated due to n=1
Statistical Analysis 1: Comparison: Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous; Test type: Superiority; p = 0.018, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; LS Mean of Difference = 6.475, 90% CI 2-sided [1.4443 to 11.5056]
Statistical Analysis 2: Comparison: Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous; Test type: Superiority; p = 0.214, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; LS Mean of Difference = 6.019, 90% CI 2-sided [-7.1464 to 19.1844]
Statistical Analysis 3: Comparison: Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous vs Cohort 2 (Day 1 - 29) Placebo for F508del Heterozygous; Test type: Superiority; p = 0.286, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; LS Mean of Difference = 7.290, 90% CI 2-sided [-15.1860 to 29.7660]

9. Secondary Outcome: Absolute Change in CF Questionnaire-Revised (CFQ-R) Respiratory Domain Score From Baseline.
Description: The CF Questionnaire-Revised (CFQ-R) Respiratory Domain Score is designed for use in participants with a diagnosis of cystic fibrosis and is designed to measure impact on overall health, daily life, perceived well-being, and symptoms. CFQ-R has a total of 50 questions. Questions 40, 41, 42, 44, 45, 46, scored 1, 2, 3, or 4, from worst to best, were used to calculate the respiratory domain score. The scaled score for the domain is calculated as 100 × (mean scores of all non-missing questions - 1) / 3, ranging from 0 to 100. If more than 3 questions in the domain have missing scores, the scaled score was set as missing. Note: The LS mean is estimated using the linear regression on the change in CFQ-R from baseline to day 29. The higher CFQ-R respiratory score indicates better health. A positive change in CFQ-R respiratory score since baseline indicates improved health quality, while a negative change indicates a decreased health quality.
Time Frame: Day 1 (Baseline) through Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous | Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous | Cohort 2 (Day 1 - 29) Placebo for F508del Heterozygous | Cohort 3 (Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Homozygous | Cohort 3(Day 1 - 29)Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Heterozygous
Number analyzed (Participants) | 19 | 7 | 4 | 3 | 1
score on a scale | 5.56 (15.930) | 10.32 (19.092) | -5.56 (21.754) | -9.26 (22.453) | -22.22 (NA) — value could not be estimated due to n=1
Statistical Analysis 1: Comparison: Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous; Test type: Superiority; p = 0.057, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; LS Mean of Difference = 5.6, 90% CI 2-sided [-0.26 to 11.37]
Statistical Analysis 2: Comparison: Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous; Test type: Superiority; p = 0.088, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; LS Mean of Difference = 8.6, 90% CI 2-sided [-2.18 to 19.40]
Statistical Analysis 3: Comparison: Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous vs Cohort 2 (Day 1 - 29) Placebo for F508del Heterozygous; Test type: Superiority; p = 0.142, Mixed Models Analysis — One-sided p-value; p-value <=0.05 indicates significance; Note: The LS mean is estimated using the linear regression on the change in CFQ-R from baseline to day 29; LS Mean of Difference = 11.2, 90% CI 2-sided [-6.90 to 29.25]

10. Secondary Outcome: Cohort 3: Absolute Change From Baseline Through Day 29 in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: as for outcome 6
Time Frame: Day 1 (Baseline) through Day 29
Population: as for outcome 1
Measure: Mean (Full Range); unit: % ppFEV1
Groups:
- Cohort 3 (Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Heterozygous: F508del Heterozygous CF participants received Galicaftor/nNavocaftor/ABBV-576 triple combination therapy (Day 1 - 29).
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
  ABBV-576: 5 mg QD, Oral capsules
Arm/Group | Cohort 3 (Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Homozygous | Cohort 3 (Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Heterozygous
Number analyzed (Participants) | 3 | 1
% ppFEV1 | -5.7 [-9.0 to -3.0] | -9.0 [-9.0 to -9.0]

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment to the end of study, median time on follow up in Part 1 was 28 days (d) for Cohort 1 (C1). In Part 2, was 28d for C1; 28 and 28d for C2; and 14, 20.5, and 14d for C3. Treatment-emergent AEs and serious AEs were collected from first dose of study drug until 30d after the last dose of study drug; mean duration on study drug in Part 1 was 28.2d for C1. In Part 2, was 25.8d for C1; 28 and 28.3d for C2; and 16.8, 20.5, and 17.5d for C3.
Description: For Cohort 1 - Triple Combination Treatment arm, a TEAE was collected through day 56 and within 30 days after the last dose of study drug.
Groups:
- Cohort 1 (Day -29 to -1) Dual Combination Galicaftor + Navocaftor for F508del Homozygous: F508del Homozygous cystic fibrosis (CF) participants received Galicaftor/Navocaftor dual combination (Day
  -29 to -1).
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
- Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous: F508del homozygous CF participants from Cohort 1(Day -29 to -1) who received Galicaftor/ Navocaftor dual combination therapy.
  followed by
  Galicaftor/Navocaftor/ABBV-119 triple combination therapy (Day 1- 29).
  Galicaftor: 300 mg QD, Oral capsules
  Navocaftor: 50 mg QD, Oral capsules
  ABBV-119: 210 mg BID, Oral capsules
Arm/Group | Cohort 1 (Day -29 to -1) Dual Combination Galicaftor + Navocaftor for F508del Homozygous | Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous | Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous | Cohort 2 (Day 1 - 29) Placebo F508del Heterozygous | Cohort 3 (Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Homozygous | Cohort 3(Day 1 - 29)Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Heterozygous
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/9 | 0/4 | 0/9 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/24 | 0/9 | 0/4 | 1/9 | 0/2
Other Adverse Events (participants affected / at risk) | 4/24 | 10/24 | 4/9 | 2/4 | 7/9 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Day -29 to -1) Dual Combination Galicaftor + Navocaftor for F508del Homozygous (N=24) | Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous (N=24) | Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous (N=9) | Cohort 2 (Day 1 - 29) Placebo F508del Heterozygous (N=4) | Cohort 3 (Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Homozygous (N=9) | Cohort 3(Day 1 - 29)Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Heterozygous (N=2)
CYSTIC FIBROSIS (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFECTIVE EXACERBATION OF BRONCHIECTASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Day -29 to -1) Dual Combination Galicaftor + Navocaftor for F508del Homozygous (N=24) | Cohort 1(Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-119 for F508del Homozygous (N=24) | Cohort 2(Day 1 - 29) Triple Combination Galicaftor+ Navocaftor + ABBV-119 for F508del Heterozygous (N=9) | Cohort 2 (Day 1 - 29) Placebo F508del Heterozygous (N=4) | Cohort 3 (Day 1 - 29) Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Homozygous (N=9) | Cohort 3(Day 1 - 29)Triple Combination Galicaftor + Navocaftor + ABBV-576 for F508del Heterozygous (N=2)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DISTAL INTESTINAL OBSTRUCTION SYNDROME (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
STEATORRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHEST DISCOMFORT (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFECTIVE PULMONARY EXACERBATION OF CYSTIC FIBROSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NASAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FORCED EXPIRATORY VOLUME DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FORCED VITAL CAPACITY DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SPIROMETRY ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 2 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POST-TRAUMATIC HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CATARRH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (5) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPUTUM INCREASED (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT04853368/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/68/NCT04853368/SAP_001.pdf